CLINICAL TRIAL: NCT04151056
Title: Impact of the Social Determinants of Health in the Central Catalan Region
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Collaborators: Institut Català de la Salut (Other)
Responsible Party: Sponsor
Other Study IDs: 19/079-P
Record Dates: First submitted 2019-10-31; First posted 2019-11-05 (Actual); Last update posted 2020-06-23 (Actual); Status verified 2019-07

CONDITIONS: Social Determinants of Health; Primary Health Care
Keywords: social determinants of health, reporting socials problems

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Patients without social determinant of health: Patients without any of the five selected social determinants of health / Patients without any of the five selected social diagnosis. Patient with a registered diagnostic " Health check" (Z00.00)
- Patients with the social determinant"stressful work hours": Patients with the selected social determinant of health. Patients with a registered diagnostic "stressful work hours " (Z56.3)
- Patients with the social determinant of health "living alone": Patients with the select social determinant of health . Patients with the selected social determinant of health . Patients with a registered diagnostic " living alone problems" (Z60.2)
- Patients with the social determinant of health "acculturation": Patients with the selected social determinant of health. Patients with a registered diagnostic "difficulty acculturation " (Z60.3)
- Patients with the social determinant "near surrounding": Patients with the selected social determinant of health. Patients with a registered diagnostic "other specific problems related to the nearest surroundings" (Z63.8)
- Patients with the social determinant "unemployment": Patients with the selected social determinant of health. Patients with a registered diagnostic "unemployment not specified" (Z56.0)

SUMMARY:
The objective of this study is to increase the registry of social determinants of health in the primary care centers and evaluate the relationship that these social determinants of health with various variables of social impact.

DETAILED DESCRIPTION:
Currently, the social problems are hidden behind clinical diagnostics. This may lead to overdiagnosis and overtreatment of some discomforts/pathologies that are observed in primary care centers that may respond better to community level interventions and promotion of health actions.

It is longitudinal , multicentered, pre and post intervention study, conducted by health professionals of central Catalonia sanitary region during 2019 Prior to the intervention, the number and type of social coded diagnoses in the clinical history is going to be described. Subsequently, an intervention will be carried out: training the professionals in the homogeneous codification of five selected social determinants. This codification will be systematically applied .The number and type of social diagnostics registered in the pre and post-intervention periods is going to be compared. Finally, the impact analysis of the social determinants is going to be carried out.

Afterwards the investigators plan to search solutions at Community level for the select social diagnoses

ELIGIBILITY:
Inclusion Criteria:

Phase I:

* Patients have been attended in their primary care centers during 23 September 2019 to 23 April 2020.
* The health professionals should complete the study checklist for each patient .

Phase II:

•Patients should sign the informed consent form to enter in a study cohort.

Exclusion Criteria:

Patients with advanced cognitive impairment because they would not be able to complete the study checklist. The study checklist is consist in answering five questions.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Study population: Population assigned and attended at the 32 centers of primary care centers from the Catalan health institute of the Central Catalonia Sanitary Region.
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2019-09-23 (Actual); Primary Completion 2021-05-23 (Estimated); Study Completion 2021-07-23 (Estimated)

PRIMARY OUTCOMES:
Population Taxes | 12 month
  In the descriptive basal analysis, the population taxes of all social diagnoses is going to be described.

SECONDARY OUTCOMES:
Sociodemographic subcategories | 7 month
  The sociodemographic data described in the study are:
  * age;
  * sex;
  * primary care team where the patient is visited;
  * type of primary care team (rural/urban);
  * index Aquas of deprivation ;
  * professional situation;
  * cultural origin of the person;
  * if cultural origin is not Spanish, years of residence in the country.
Comparison with the post-intervention data of the six diagnostics with Chi Quadrat Test. | 7 month
  For this comparison is going to be used independent samples in the different subcategories.
  The 6 diagnostics used are:
  * health check;
  * stressful work hours;
  * living alone problems ;
  * difficult acculturation
  * other specific problems related to the nearest surrounding;
  * unemployment not specified.
Social Impact. Parametric and non parametric test | 12 month
  It will be evaluated health differences in the six coded groups (including the control group) through appropriate parametric and non-parametric tests , It is going to be compared the average of each selected dependent health variables in social coded diagnoses and the screened patients group without a social diagnosis
  The dependent health variables are going to be analysed after the codification of the six selected diagnosis. The study dependent health variables are:
  * number of clinical diagnoses registered;
  * number of medicines consumed ;
  * number of the total diagnostic test requested;
  * number of specialists referrals
  * number of visits to health centers

CONTACTS AND LOCATIONS:
Overall Officials: Jacobo Mendioroz peña, MD, Study Chair — Institut Català de la Salut
Locations (1):
- Primary healthcare consultations of the Catalan health institute of the central catalonia region, Manresa, Barcelona, Spain

REFERENCES:
- [Derived] Rodoreda-Pallas B, Lumillo-Gutierrez I, Miro Catalina Q, Torra Escarrer E, Sanahuja Juncadella J, Morin Fraile V. Recording of Social Determinants in Computerized Medical Records in Primary Care Consultations: Quasi-Experimental Study. JMIR Form Res. 2023 Jan 25;7:e41706. doi: 10.2196/41706. PMID 36696168